CLINICAL TRIAL: NCT03483233
Title: Neural Bases of the Check Process
Acronym: Check
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0143; 2018-A00405-50 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-03-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Gyrus Cinguli; Cognitive Control Process; Check process; Decision Making; fMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI and EEG study (Experimental)
  Interventions: Other: fMRI and EEG study

INTERVENTIONS:
Other: fMRI and EEG study — fMRI and EEG study

SUMMARY:
Effective exploration of the environment, check for information to improve one's own performance, are fundamental abilities of human cognition. These abilities are dependent on the process of cognitive control.

However, they are clearly impaired and uncontrollable in certain behavioral disorders such as obsessive-compulsive disorder (OCD). Compulsive checks of these patients, spontaneously associated with a feeling of intense uncertainty, suggest disturbances of evaluative and metacognitive functions. However, no biological observations have yet been able to feed these hypotheses.

The evaluation of decisions and actions involves the middle cingulate cortex (MCC) (which belongs to a cortico-subcortical network structurally and functionally altered in OCD patients). Cingulotomy has long been used as a therapy in severe OCD, with However, the precise part of the cingulate cortex that contributes to check (and its pathological forms) remains to be discovered.

The purpose of this research campaign is to determine, through functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) in healthy human subjects:

1. the location and role of the MCC region involved in normal check decision processes,
2. determine the identity of the entire network involved

ELIGIBILITY:
Inclusion Criteria:

* adults age range 20-45 years
* being able to provide a written consent form
* having a social insurance
* have a normal vision (with or without corrections)
* Right-handed

Exclusion Criteria:

* Subjects with MRI contraindications (e.g. pacemaker, claustrophobia, metal in the body, etc…).
* Pregnant subjects
* Subjects with neurological history
* Subjects must be willing to be advise in case of discovery of brain abnormality.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Measuring changes in brain activity in regions of interest when performing cognitive tasks. | through study completion, an average of 3 years
  Behavior: Measurement of reaction times of correct answer during cognitive task.
  fMRI and EEG: Brain activity signal,
Measuring changes in brain activity in regions of interest when performing cognitive tasks. | through study completion, an average of 3 years
  Behavior: Measurement of % of correct answer during cognitive task.
Measuring changes in brain activity in regions of interest when performing cognitive tasks. | through study completion, an average of 3 years
  - Measurement of the amplitude of the BOLD signal change in MRI according to the different cognitive tasks in the different regions of interest. Measurement of resting GABA and Glutamate concentrations in the different regions of interest.
  Measurement of the amplitude of the change of the electrical signal in EEG according to the different cognitive tasks in the different regions of interest.

SECONDARY OUTCOMES:
Calculation of the correlations in the regions of interest of the individual values of the Blood Oxygen Level Dependent (BOLD) signal with the data of the concentration of Acide γ-aminobutyrique (GABA) | through study completion, an average of 3 years
  calculate with the bold signal (spectroscopy)
Calculation of the correlations in the regions of interest of the individual values of the Blood Oxygen Level Dependent (BOLD) signal with the data of the amplitude of the electrical signal (EEG) | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Procyk, Principal Investigator — INSERM U1208
Locations (1):
- Inserm U1208, Bron, France

REFERENCES:
- [Result] Stoll FM, Fontanier V, Procyk E. Specific frontal neural dynamics contribute to decisions to check. Nat Commun. 2016 Jun 20;7:11990. doi: 10.1038/ncomms11990. PMID 27319361